CLINICAL TRIAL: NCT03962049
Title: Evaluation of the Safety and Pharmacokinetics of a Single Dose of Linzagolix in Female Subjects With Normal and Impaired Hepatic Function
Brief Title: Safety and Pharmacokinetics Study of Linzagolix in Female Subjects With Normal and Impaired Hepatic Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ObsEva SA (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 18-OBE2109-009
Record Dates: First submitted 2019-05-22; First posted 2019-05-23 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Hepatic Impairment; Healthy Participants
Keywords: Linzagolix; OBE2109; Hepatic Impairment; Hepatic Insufficiency; Liver Diseases; Clinical pharmacology study
MeSH Terms: conditions — Hepatic Insufficiency; Liver Diseases | interventions — linzagolix

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Normal Hepatic Function (Experimental): Healthy participants with Normal Hepatic Function
  Interventions: Drug: Linzagolix
- Mild Hepatic Impairment (Experimental): Presence of Mild Hepatic Impairment (score of 5 to 6, on the Child Pugh scale and with features of cirrhosis due to any etiology)
  Interventions: Drug: Linzagolix
- Moderate Hepatic Impairment (Experimental): Presence of Moderate Hepatic Impairment (score of 7 to 9, on the Child Pugh scale and with features of cirrhosis due to any etiology)
  Interventions: Drug: Linzagolix
- Severe Hepatic Impairment (Experimental): Presence of Severe Hepatic Impairment (score of 10 to 15 on the Child Pugh scale and with features of cirrhosis due to any etiology)
  Interventions: Drug: Linzagolix

INTERVENTIONS:
Drug: Linzagolix — A single dose of 200 mg linzagolix (2 tablets of 100 mg) will be administered orally under fasting conditions

SUMMARY:
The primary objective of this study is to assess the pharmacokinetics (PK) of linzagolix in subjects with varying degrees of impaired hepatic function compared to match control subjects with normal hepatic function

DETAILED DESCRIPTION:
This is a Phase 1, non-randomized, open label, single-dose study to evaluate the effect of varying degrees of impaired hepatic function (i.e., mild, moderate, and severe Hepatic Impairment (HI)) on the PK, safety, and tolerability of linzagolix and its major metabolite, KP017.

Up to 28 adult female participants will be enrolled.

ELIGIBILITY:
Key Inclusion Criteria:

Hepatic Impaired Subjects

1. Adult female, 18-75 years of age, inclusive, at screening
2. Has a BMI ≥ 18.0 and ≤ 42.0 kg/m^2 and weight ≥ 40 kg, at screening
3. Aside from HI, be sufficiently healthy for study participation based upon medical history, physical examination, vital signs, electrocardiograms (ECGs), and screening clinical laboratory profiles, as deemed by the Principal Investigator (PI) or designee
4. Has a score on the Child-Pugh scale at screening as follows:

   * Severe HI: ≥ 10 and ≤ 15
   * Moderate HI: ≥ 7 and ≤ 9
   * Mild HI: ≥ 5 and ≤ 6
5. Has a diagnosis of chronic (> 6 months), stable (no acute episodes of illness within the previous 2 months due to deterioration in hepatic function) hepatic insufficiency with features of cirrhosis due to any etiology

Healthy Subjects

1. Healthy adult female will be matched based upon age and BMI
2. Medically healthy with no clinically significant medical history, physical examination, laboratory profiles, vital signs or ECGs, as deemed by the PI or designee.

Key Exclusion Criteria:

Hepatic Impaired Subjects

1. Has a clinically active Grade 3 or 4 encephalopathy
2. Has fluctuating or rapidly deteriorating hepatic function within the screening period, and up to 30 days prior to Day 1, in the opinion of the PI and Sponsor
3. Has history of liver or other solid organ transplant
4. Had any major surgery within 4 weeks prior to dosing
5. Has a surgical (e.g., hepatectomy, nephrectomy, digestive organ resection) or medical condition other than HI which might significantly alter the absorption, distribution, metabolism, or excretion of linzagolix and its metabolites, or which may jeopardize the subject's safety in case of participation in the study in the opinion of the PI or designee

Healthy Subjects

1. Has any clinically significant illness, as judged by the PI or designee, within 4 weeks prior to dosing
2. Has laboratory values at screening or check-in which are deemed to be clinically significant (especially derangement within liver function test), unless agreed in advance by the PI and the Sponsor

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2019-05-15 (Actual); Primary Completion 2019-10-23 (Actual); Study Completion 2019-11-01 (Actual)

PRIMARY OUTCOMES:
Plasma pharmacokinetic (PK) parameter Cmax of linzagolix and of KP017 | predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120 hours post-dose
  Measurement of effect of hepatic impairment on PK of linzagolix and its metabolite KP017 by assessment of the maximum plasma concentration (Cmax). Cmax directly determined from the plasma concentration-time profiles
Plasma PK parameter Tmax of linzagolix and of KP017 | predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120 hours post-dose
  Measurement of effect of hepatic impairment on PK of linzagolix and its metabolite KP017 by assessment of the Time to reach Cmax (Tmax)
Plasma PK parameter AUC0-t of linzagolix and of KP017 | predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120 hours post-dose
  Measurement of effect of hepatic impairment on PK of linzagolix and its metabolite KP017 by assessment of the AUC0-t (area under the concentration time curve, from time 0 to the last observed non-zero concentration)
Plasma PK parameter T1/2 of linzagolix and of KP017 | predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120 hours post-dose
  Measurement of effect of hepatic impairment on PK of linzagolix and its metabolite KP017 by assessment of the T1/2 (Terminal half life)

SECONDARY OUTCOMES:
Treatment emergent Adverse Events | Day 1 to 14 days post-dose
  Assessment of safety and tolerability of a single dose of linzagolix in hepatic impaired subjects compared with healthy control subjects by assessing the number, frequency and severity of treatment emergent Adverse Events

CONTACTS AND LOCATIONS:
Overall Officials: ObsEva SA, Study Director — Geneva
Locations (2):
- United States (2):
  - Clinical Site, Hialeah, Florida
  - Clinical Site, Orlando, Florida